CLINICAL TRIAL: NCT07177573
Title: The Effects of Virtual Reality on Pain, Anxiety, and Comfort During Continuous Passive Motion After Total Knee Arthroplasty
Brief Title: Virtual Reality During Passive Motion After Knee Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Emel Yılmaz, Professor, Manisa Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCBU-SBF-EY-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Virtual Reality; Continuous Passive Movement Therapy; Pain; Anxiety; Comfort; Patient
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Virtual Reality
  Interventions: Other: Virtual Reality
- Control (No Intervention)

INTERVENTIONS:
Other: Virtual Reality — The demographic information of the participants will be collected through face-to-face interviews. Pain and comfort levels will be assessed using the Visual Analog Scale (VAS) prior to the intervention. Additionally, anxiety levels will be measured with the Spielberger State-Trait Anxiety Inventory, and vital signs will be recorded. Patients included in the study will be informed about the use of virtual reality (VR) goggles and introduced to the videos that will be viewed. During the Continuous Passive Motion (CPM) application, patients will be positioned in a semi-Fowler's position with a pillow placed under the head for support. Through virtual reality, patients will watch the video Forest Walk along the Middle Fork Snoqualmie River Trail with Relaxing Sounds and the accompanying sounds will be delivered through headphones integrated into the goggles.
  Arms: Experimental

SUMMARY:
The purpose of this study is to investigate the effects of virtual reality on pain, anxiety, and comfort during continuous passive motion following total knee arthroplasty

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of virtual reality on pain, anxiety, and comfort during continuous passive motion following total knee arthroplasty Study Hypotheses

H0: The use of virtual reality during continuous passive motion following total knee arthroplasty does not reduce pain levels.

H1: The use of virtual reality during continuous passive motion following total knee arthroplasty reduces pain levels.

H0: The use of virtual reality during continuous passive motion following total knee arthroplasty does not reduce anxiety levels.

H1: The use of virtual reality during continuous passive motion following total knee arthroplasty reduces anxiety levels.

H0: The use of virtual reality during continuous passive motion following total knee arthroplasty does not improve comfort levels.

H1: The use of virtual reality during continuous passive motion following total knee arthroplasty improves comfort levels.

Study Population and Sample Size

The study population will consist of patients undergoing total knee arthroplasty at the Orthopedics and Traumatology Department of Manisa Celal Bayar University Hafsa Sultan Hospital between August 2025 and August 2026. The sample size was calculated using G*Power 3.1. Assuming a moderate effect size (d = 0.5) for the differences between intervention and control groups regarding postoperative pain and comfort levels, with 80% power and α = 0.05, the minimum sample size required is 102 patients (n1 = 51, n2 = 51).

Inclusion Criteria

* First-time total knee arthroplasty
* Postoperative day 2
* Mobilized before CPM application
* Adequate vision and hearing to use the virtual reality device
* Oriented to person, place, and time
* No cognitive, sensory, or verbal communication impairments
* No history of vertigo
* No hypertension
* Not using sedative, anxiolytic, or similar medications
* Willing to voluntarily participate in the study

Exclusion Criteria

* Any diagnosed psychiatric disorder
* History of vertigo
* Hypertension
* Using sedative, anxiolytic, or similar medications
* Poor general condition
* Unwillingness to participate Randomization

The study will include 102 patients meeting the eligibility criteria, providing written informed consent, and completing pretests. Patients will be randomized into the virtual reality group or control group using a computer-generated program to ensure allocation concealment and minimize bias (https://www.randomizer.org

). Block randomization will be applied with equal distribution between groups. At the start of the study, opaque sealed envelopes will designate which letter corresponds to each group: A for the virtual reality group and B for the control group. Numbered blocks from the randomization list will be placed in a black bag. Each incoming patient will be assigned to a group based on the block drawn from the bag. The process will continue until all blocks are assigned.

To ensure transparency, completeness, and clarity in reporting, all stages of this randomized controlled trial will follow the CONSORT 2010 guidelines.

Dependent and Independent Variables

Dependent Variables: Patients' state anxiety scores, pain scores, and comfort scores.

Independent Variable: Virtual reality intervention.

Control Variables: Patients' age, gender, education level, occupation, marital status, prior surgical experience, knowledge about virtual reality, and similar demographic and clinical factors.

Data Collection Instruments

The following instruments will be used to collect study data:

Personal Information Form:

A form developed by the researchers to assess patients' age, gender, education level, occupation, marital status, previous surgical experiences, and knowledge about virtual reality.

Visual Analog Scale (VAS):

The VAS is a unidimensional scale widely accepted for assessing acute and chronic pain intensity. It is reliable, simple, and easy to use. The scale ranges from 0 ("no pain") to 10 ("extremely severe pain"). In this study, the VAS will be used to evaluate both pain and comfort levels.

State-Trait Anxiety Inventory (STAI):

The STAI is a self-report questionnaire consisting of short statements, rated on a 4-point Likert scale. It has two subscales: the State Anxiety Scale (STAI-I) and the Trait Anxiety Scale (STAI-II), each containing 20 items.

The state anxiety subscale measures the emotional state experienced by an individual at a specific moment under certain conditions.

The trait anxiety subscale assesses how frequently an individual generally experiences anxiety in daily life.

The scale includes both direct and reverse-scored items. Direct items reflect negative emotions, while reverse-scored items indicate positive emotions. For the state anxiety subscale, reverse-scored items are: 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The total score is calculated by subtracting the sum of reverse-scored items from the sum of direct items and adding a constant value of 29. The fixed constant for the state anxiety subscale is 50. Scores range from 20 to 80, with higher scores indicating higher anxiety.

Pilot Testing To ensure the clarity, feasibility, and usability of the data collection instruments, a pilot study will be conducted with five patients meeting the study criteria and who consent to participate, admitted to the Orthopedics and Traumatology Department of Manisa Celal Bayar University Hafsa Sultan Hospital between September 1-31, 2025. Based on feedback from the pilot, necessary adjustments will be made to the data collection forms. Patients who participate in the pilot study will be excluded from the main study.

Study Procedure

Patients who have undergone total knee arthroplasty (TKA) and are scheduled for continuous passive motion (CPM) on postoperative day 2 will be identified. Eligible patients will be taken to the physiotherapy and rehabilitation room of the Orthopedics and Traumatology Department for CPM. The session for each patient will begin at 10:00 AM. CPM will be performed under the supervision of a physiotherapist, after which patients will be returned to their rooms.

Intervention Group (Virtual Reality Group)

At the start of the study, eligible patients will be informed about the study's purpose and procedures, and verbal and written informed consent will be obtained. Demographic information will be collected via face-to-face interview. Pre-intervention assessments will include:

Pain and comfort levels, measured using the Visual Analog Scale (VAS) Anxiety levels, measured using the State-Trait Anxiety Inventory (STAI) Vital signs, recorded prior to the intervention Patients will be briefed on the use of the virtual reality headset and introduced to the selected video content. During CPM, patients will be positioned in a semi-Fowler position with a pillow under the head for support.

Virtual Reality Device:

* VR Shinecon G06a Resin Lens 720° Panoramic 3D Stereo Virtual Reality --Headset (https://www.trendyol.com/vr-shinecon/g06a-recine-lens-720-panoramik-3d-stereo-sanal-gerceklik-gozlugu-metaverse-popsoket-p-239865451)
* Compatible with 3.5-6.0 inch Android and iOS smartphones
* Provides panoramic view through two equal split-screen lenses
* Does not require additional power supply or connection unit
* Ergonomic and lightweight, allowing comfortable long-term use
* Equipped with gyroscope, accelerometer, and head-tracking sensors for immersive experience

Virtual Content:

"Participants will watch a forest walking video along the Middle Fork Snoqualmie River Trail available on YouTube (https://www.youtube.com/watch?v=vlbF9imkUMM-

) with relaxing nature sounds. The video audio will be delivered through fixed headphones on the VR headset. Copyright permission for the video was obtained by subscribing and paying the fee via the website (https://4krelax.com/video/19/896459643/4k-forest-walk-along-middle-fork-snoqualmie-river-trail-hiking-with-relaxing-nature-sounds).

During the Intervention:

* Patients will watch the VR video for 20 minutes while CPM is applied
* Post-intervention, the headset will be removed, and vital signs recorded again
* All pre-intervention scales (VAS, STAI, comfort assessments) will be re-administered

Hygiene Protocol:

* A disposable eye mask will be used for each patient
* Headset surfaces will be disinfected after each use Control Group

At the start of the study, patients in the control group will be informed about the study and verbal and written consent will be obtained. Demographic information will be collected via face-to-face interview. Pre-intervention assessments will include:

Pain and comfort levels, measured using the Visual Analog Scale (VAS)

Anxiety levels, measured using the State-Trait Anxiety Inventory (STAI)

Vital signs, recorded prior to the intervention

After the CPM session, vital signs will be re-evaluated, and all pre-intervention scales (VAS, STAI, comfort assessments) will be re-administered.

Patients in the control group will receive routine care only; no additional interventions will be applied.

During the study, all devices used to measure vital signs will be pre-calibrated. Data collection will be performed by the same researcher for all participants to maintain consistency, and no additional observers will be involved. The CPM session and assessments will be repeated on postoperative day 3 following the same procedures.

Data Analysis

Data will be analyzed using SPSS version 25.0 (Statistical Package for the Social Sciences). Descriptive statistics will be presented as frequencies and percentages for categorical variables, and as mean ± standard deviation, median, minimum, and maximum values for continuous variables.

For comparisons between groups:

Categorical variables will be analyzed using Chi-square or Fisher's Exact tests.

Continuous variables with normal distribution will be compared using independent two-sample t-tests for between-group comparisons and paired t-tests for within-group comparisons over two time points.

Non-normally distributed continuous variables will be compared using the Mann-Whitney U test for two-group comparisons.

For comparisons over three or more time points:

Repeated measures ANOVA will be used for normally distributed data. Friedman test will be used for non-normally distributed data. A p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

First-time total knee arthroplasty Postoperative day 2 Mobilized before CPM application Adequate vision and hearing to use the virtual reality device Oriented to person, place, and time No cognitive, sensory, or verbal communication impairments No history of vertigo No hypertension Not using sedative, anxiolytic, or similar medications Willing to voluntarily participate in the study

Exclusion Criteria:

* Any diagnosed psychiatric disorder
* History of vertigo
* Hypertension
* Using sedative, anxiolytic, or similar medications
* Poor general condition
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain, Anxiety, and Comfort Levels during Continuous Passive Motion | Immediately before and after each CPM session on postoperative day 2 and day 3
  Pain and comfort levels will be assessed using the Visual Analog Scale (VAS, 0-10), where 0 indicates no pain/comfort and 10 indicates worst pain/maximal comfort. Anxiety will be measured using the State-Trait Anxiety Inventory (STAI). The effects of virtual reality during CPM on pain, anxiety, and comfort will be compared between the VR and control groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://4krelax.com/video/19/896459643/4k-forest-walk-along-middle-fork-snoqualmie-river-trail-hiking-with-relaxing-nature-sounds